CLINICAL TRIAL: NCT07113756
Title: Efficacy of Topical Metformin 30% Cream Versus Betamethasone Valerate 0.1% Cream in Treatment of Adult Patients With Plaque Psoriasis
Brief Title: New Topical Treatment in Plaque Psoriasis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sherein Gamal Abdellah, assistant lecturer of dermatology, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Soh-Med-25-2-2MD
Record Dates: First submitted 2025-07-23; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group (1) will use topical metformin 30% cream (Active Comparator): each patient will use topical metformin 30% cream twice daily for 12 weeks.
  o Preparation of metformin 30% cream: Weighing 30 gm standard metformin ( E. Merck ) supplied by chemtech. Using digital balance then Grinding the powder by pestle & Morter then Adding 30 ml propylene glycol and alcohol to reach a total 100 gm weight then adding parabens mix as preservative with 0.5 gm then mix thoroughly followed by Levegating & mixing then divide to smaller well tighten closure with labels
  Interventions: Drug: topical metformin 30% cream
- group(2) topical betamethasone valerate .1% cream. (Placebo Comparator): each patient will use topical betamethasone valerate .1% cream twice daily for 12 weeks.
  Interventions: Drug: betamethasone valerate.1% cream

INTERVENTIONS:
Drug: topical metformin 30% cream — each patient will use topical metformin 30% cream twice daily for 12 weeks.
  o Preparation of metformin 30% cream: Weighing 30 gm standard metformin ( E. Merck ) supplied by chemtech. Using digital balance then Grinding the powder by pestle & Morter then Adding 30 ml propylene glycol and alcohol to reach a total 100 gm weight then adding parabens mix as preservative with 0.5 gm then mix thoroughly followed by Levegating & mixing then divide to smaller well tighten closure with labels
  Arms: group (1) will use topical metformin 30% cream
Drug: betamethasone valerate.1% cream — each patient (age, sex and BMI matched) will use topical betamethasone valerate 0.1% cream twice daily for 12 weeks.
  o Manufactured by Egyptian international pharmaceutical industries co. E.I.P.I.C.O. and will be purchased from local pharmacy, Sohag, Egypt.
  Arms: group(2) topical betamethasone valerate .1% cream.

SUMMARY:
Psoriasis is a chronic, recurring, immune-mediated papulosquamous condition The etiology of psoriasis is complex and not fully understood Though many treatment options are available for plaque psoriasis, each has its limitations and side effects. Therefore, the need for an effective topical agent that delivers the drug efficiently into the target site with minimal systemic side effects remains an aim in itself.Metformin is a derivative of biguanide that is the most widely used as an oral antihyperglycemic agent for the control of diabetes mellitus. In addition to its hypoglycaemic effect, metformin can serve as an anti-inflammatory agent. Metformin has been demonstrated to suppress proliferation in keratinocytes by blocking the mitogen-activated protein kinase pathway (MAPK) (25). Hence, metformin may play an important role in the reducing pathogenesis of psoriasis by anti-inflammatory, anti-proliferative, and anti- angiogenic effects .The topical form of metformin has been used in regenerative medicine (33), treatment of acne (34), adjuvant treatment for psoriasis (35), neo-adjuvant therapy for squamous cell carcinoma (36), and treatment of pigmentary disorders as an alternative to hydroquinone (37). The aim of the study is to:

* Assess the efficacy and the safety of topical metformin 30% cream compared with betamethasone valerate 0.1 % cream in the treatment of adult patients with mild and moderate plaque psoriasis.
* Compare the efficacy of topical metformin 30% cream versus betamethasone valerate 0.1 % cream clinically, dermoscopically, histopathologically and immunohistochemically by measuring tissue level of IL17 in psoriatic skin lesions before and after treatment in all patients.

ELIGIBILITY:
* Inclusion Criteria:

  * Patients of both sexes aged ≥ 18 years, having clinical and dermoscopic finding of mild and moderate plaque psoriasis and did not receive any topical, phototherapy or systemic treatment in the last 3 months for psoriasis.
* Exclusion Criteria:

  * Other types of psoriasis
  * Patient refusal.
  * Pregnant and lactating women.
  * Patients with other inflammatory or autoimmune skin diseases (atopic dermatitis, lichen planus, alopecia areata, cutaneous lupus erythromatosis, systemic sclerosis, rheumatoid arthritis, acne vulgaris, hidradinitis supprativa
  * Hypersensitivity to topical treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
clinical improvement in psoriatic skin lesions | at the end of treatment (12 weeks) and 3 months after stoppage of treatment
  clinical evaluation using PASI score to assess improvement before and treatment

CONTACTS AND LOCATIONS:
Overall Officials: shereen G gamal, Assistant lecturer, Principal Investigator — Sohag University

IPD SHARING:
Plan to Share IPD: No
individual participant data will not be shared due to patient privacy concerns and lack of consent for external sharing